CLINICAL TRIAL: NCT02973698
Title: Effects of a Speech-Language Pathology Intervention on Individuals With Parkinson's Disease
Brief Title: Benefit From the Chin Down Maneuver in the Swallowing Performance and Self-perception of Parkinson's Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 140263
Record Dates: First submitted 2016-11-22; First posted 2016-11-25 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Dysphagia, Oropharyngeal; Parkinson Disease; Speech Therapy; Orientation
MeSH Terms: conditions — Deglutition Disorders; Parkinson Disease; Communication Disorders; Orientation, Spatial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- chin-down posture maneuver (Other): The patients in received an intervention program consisting of four weekly individual sessions of 30 minutes. In these sessions, it was performed the training of Chin-down postural maneuver with saliva and water. The participants were trained to perform the maneuver twice a day, swallowing saliva, and during meals, throughout the week, at home. The participants received a form, so they recorded the number of times they performed the maneuver at home. It allowed the control of adherence, being reinforced at each session the importance of adherence to treatment. Besides, the subjects received instructions regarding feeding. All the instructions, as well as the explanation about the maneuver, were submitted to the patients through a written document.
  Interventions: Other: chin-down posture maneuver; Other: Orientations about swallowing
- Control (Other): The participants of this group underwent evaluation of swallowing, and the same assessment was repeated after four weeks, without any intervention during that period.
  Interventions: Other: Control
- Orientations about swallowing (Other): The individuals participated in an intervention program which consisted of four individual sessions a week, with 30 minutes. In these sessions, the instructions about feeding were performed. The individuals received all the instructions on a written document. In the sessions, it was verified doubts about the guidelines and treatment adherence. In this group, it was not applied the Chin-down postural maneuver.
  Interventions: Other: Orientations about swallowing

INTERVENTIONS:
Other: chin-down posture maneuver — it was performed the training of Chin-down postural maneuver with saliva and water. Besides, the subjects received instructions regarding feeding.
  Arms: chin-down posture maneuver
Other: Orientations about swallowing — The instructions about feeding were performed. The individuals received all the instructions on a written document.
  Arms: Orientations about swallowing; chin-down posture maneuver
Other: Control — No intervention will do
  Arms: Control

SUMMARY:
Objective: To verify the effectiveness of chin-down posture maneuver in swallowing therapy for Parkinson's disease (PD).

DETAILED DESCRIPTION:
Participants Participants were PD patients recruited from a Parkinson´s disease and Movement Disorders Clinic from Hospital de Clínicas de Porto Alegre (HCPA), a reference hospital, in the Rio Grande do Sul, Brazil. It was obtained from participants the written free and informed consent to participate in the research. This study was approved by the hospital central research ethics committee.

Inclusion and exclusion criteria Patient evaluation It was performed cognitive screening which consists of Mini-Mental State Examination (MMSE) and Montreal Cognitive Assessment (MoCA) in all patients before the intervention. It was also applied the instruments Parkinson Disease Questionnaire-39 (PDQ-39), translated to Portuguese, and the Beck Depression Inventory (BDI). These tests were applied to verify the influence of cognitive aspects, depression and quality of life in the therapeutic process.

To evaluate the intervention's effectiveness, an evaluation of swallowing was conducted in two moments (before and after intervention). Three kinds of assessments were performed: (1). Fiberoptic endoscopic evaluation of swallowing (FEES); (2) Clinical evaluation and (3) assessment of the quality of life related to swallowing (SWALQOL).

* Fiberoptic endoscopic evaluation of swallowing (FEES): This objective examination of swallowing was performed according to the following protocol: First, it was tested the prior state of secretion in the nasopharyngeal structures, oropharynx, and laryngopharynx. Next, the individual received liquid consistency offered through a syringe, 3 and 5ml of water with edible blue food coloring. For the pasty consistency, 3 and 5ml of thickened water were provided through a syringe with edible blue food coloring. It was offered ¼- water and salt biscuits with good blue food coloring to assess the solid consistency. No anesthetic was used for the examination. The images were later analyzed by an otolaryngologist physician, experienced in the dysphagia area. It was observed the presence of thickening on the posterior laryngeal wall, tremor in structures (base of tongue and vallecula), early escape (characterized by the presence of food in the hypopharynx or larynx before the swallowing reflex was triggered), vallecular stasis in glossoepiglottic folds and pyriform sinus (characterized by accumulation of food after the third swallowing on the mentioned structures), penetration (characterized by the presence of food in the laryngeal vestibule), tracheal aspiration (characterized by food intake in the region located below the vocal folds, in the subglottic region and in the trachea, at any time of swallowing) and cough reflex. The alterations were classified as present or absent. The equipment used was the flexible nasopharyngoscope Maschida ENT-III, 3.2mm, with Xerônio Storz light source.
* Clinical evaluation and Functional Oral Intake Scale (FOIS): clinical evaluation of swallowing was performed by a certified speech therapist, previously trained to apply the protocols. All the evaluations were conducted by the same professional. This assessment had the purpose of checking signs and symptoms of oropharyngeal dysphagia. It was used solid food consistency (half portion of bread) and liquid (100ml of water) evaluated by free demand. The analyzed signs and symptoms were: history of aspiration pneumonia; alert state; interaction attention/ability; awareness of the swallowing problem; awareness of secretion; ability to manipulate flows; postural control; fatigability; anatomy and oral, pharyngeal and laryngeal physiology; orofacial tonus; oral apraxia; orofacial sensitivity; gag pharyngeal contraction; saliva swallowing; cough and hawk; swallowing apraxia; oral residue; delayed swallowing reflex; reduction in laryngeal elevation; wet voice; and multiple swallowing. A total of 21 signs and symptoms were evaluated as present or absent. At the end of the objective and clinical evaluation, the intake of food was scored according to Functional Oral Intake Scale (FOIS). This scale scores the level of oral food intake of patients at specific levels, from 0 (restricted to alternative food pathway) to 7 (total oral intake with no restrictions), with the aim of monitoring the patients' evolution during the therapeutic process. A translated and validated version for Brazilian Portuguese was used.
* The quality of Life in Swallowing Disorders: The questionnaire Quality of Life in Swallowing Disorders (SWAL-QOL) was applied, to verify the symptoms presented by the patients, as well as their influence on the quality of life. This instrument has Alpha Cronbach coefficient higher than 0.80, except in one domain. Thus, it presents excellent internal consistency and short-term reproducibility. It is a sensitive scale to differentiate oropharyngeal dysphagia degrees of severity. The version translated and validated for Brazilian Portuguese was used. All questionnaires were applied in a waiting room. The questions and possible answers were read by the researcher for all patients. The questionnaires application was performed individually, for each patient.

Intervention Individuals who agreed to participate in this study were allocated to one of the three interventions groups: (1) experimental group (patients performed the chin-down posture maneuver), (2) control group (PD individuals without any intervention) and (3) orientation group (PD participants that received swallowing orientations).

1. Experimental group (EG) (chin-down posture maneuver group): patients in received an intervention program consisting of four weekly individual sessions of 30 minutes. In these sessions, it was performed the training of Chin-down postural maneuver with saliva and water. The participants were trained to perform the maneuver twice a day, swallowing saliva, and during meals, throughout the week, at home. The participants received a form, so they recorded the number of times they performed the maneuver at home. It allowed the control of adherence, being reinforced at each session the importance of adherence to treatment. Besides, the subjects received instructions regarding feeding. All the instructions, as well as the explanation about the maneuver, were submitted to the patients through a written document.
2. Control group (CG) (PD individuals without any intervention): The participants of this group underwent evaluation of swallowing, and the same assessment was repeated after four weeks, without any intervention during that period.
3. Orientations group (OG): the individuals participated in an intervention program which consisted of four individual sessions a week, with 30 minutes. In these sessions, the instructions about feeding were performed. The individuals received all the instructions on a written document. In the sessions, it was verified doubts about the guidelines and treatment adherence. In this group, it was not applied the Chin-down postural maneuver.

The EG and OG interventions were used by the same researcher, previously trained. After the end of the research, it was offered to the CG and OG individuals the same swallowing therapy performed to the GE.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Parkinson's disease and diagnosis of oropharyngeal dysphagia

Exclusion Criteria:

* presenting language and hearing disorders, which could complicate the understanding of an intervention program, diagnosis of dementia or other neurological illnesses.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-06; Primary Completion 2015-01 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Clinical evaluation of swallowing | Four weeks
  This assessment had the purpose of checking signs and symptoms of oropharyngeal dysphagia. It was used solid food consistency (half portion of bread) and liquid (100ml of water) evaluated by free demand. A total of 21 signs and symptoms were evaluated as present or absent

SECONDARY OUTCOMES:
Fiberoptic endoscopic evaluation of swallowing | Four weeks
  This objective examination of swallowing was performed according to the following protocol: First, it was tested the prior state of secretion in the nasopharyngeal structures, oropharynx, and laryngopharynx. Next, the individual received liquid consistency offered through a syringe, 3 and 5ml of water with edible blue food coloring. For the pasty consistency, 3 and 5ml of thickened water were provided through a syringe with edible blue food coloring. It was offered ¼- water and salt biscuits with good blue food coloring to assess the solid consistency.
The quality of Life in Swallowing Disorders | Four weeks
  The questionnaire Quality of Life in Swallowing Disorders (SWAL-QOL) was applied, to verify the symptoms presented by the patients, as well as their influence on the quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Maira Olchik, Principal Investigator — Hospital de Clínicas de Porto Alegre

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ayres A, Jotz GP, Rieder CR, Olchik MR. Benefit from the Chin-Down Maneuver in the Swallowing Performance and Self-Perception of Parkinson's Disease Patients. Parkinsons Dis. 2017;2017:7460343. doi: 10.1155/2017/7460343. Epub 2017 Jan 19. PMID 28203475